CLINICAL TRIAL: NCT05553288
Title: Determining the Effectiveness of a Real Time Data Safety Study Tool for Clinical Research Subjects
Brief Title: Effectiveness of a Real Time Data Safety Study Tool
Acronym: RTD
Status: Completed | Type: Observational
Sponsor: Perseverance Research Center, LLC (Other)
Collaborators: HDC (Unknown)
Responsible Party: Sponsor
Other Study IDs: RTD-01
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Study Subjects Currently Enrolled in a Clinical Research Trial
Keywords: text messaging, safety, real time data

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- active group: Every study participant will actively receive daily text messages asking about their change in health and concomitant medication.

SUMMARY:
Study RTD-01 is a non-interventional, pilot study designed to determine if a specific coded SMS text message study tool is effective in collecting daily real time safety data in subjects participating in clinical trials.

DETAILED DESCRIPTION:
This study is to determine if a daily SMS text message study tool will improve adverse event and concomitant medication reporting. Patient reported adverse events and changes in concomitant medications are essential in clinical trials to determine drug-related symptoms and side effects. This study will help identify the benefits and challenges of real time daily reported outcome measures that can later be implemented in future clinical trials to enhance trial outcomes. In addition, data collected from this study will support a more sophisticated safety study tool for future study participants.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 age inclusive
* Male or Female
* Currently enrolled in an ongoing clinical trial
* Capable of providing informed consent and complying with daily study procedures
* Must be able to receive and respond to text messages through phone provider

Exclusion Criteria:

* Subjects not currently involved in a clinical trial
* Subjects who cannot receive text messages
* Unable to comply to the study protocol and study visits

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: -Men and women from 18-85 years of age inclusive, who are currently enrolled in a clinical trial at Perseverance Research Center. All subjects must meet all inclusion and no exclusion criteria to be eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
To improve AE and concomitant medication reporting | 6 weeks
  Data collected daily through secure text messaging

SECONDARY OUTCOMES:
Decrease recall bias | 6 weeks
  Daily reporting of AEs and concomitant medication changes

CONTACTS AND LOCATIONS:
Locations (1):
- Perseverance Research Center, LLC, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No